CLINICAL TRIAL: NCT03034135
Title: A Phase II, Multicenter, Open-Label, Single-Arm Study to Evaluate the Safety, Tolerability, and Efficacy of DIsulfiram and Copper Gluconate in Recurrent Glioblastoma
Brief Title: Safety, Tolerability and Efficacy of Disulfiram and Copper Gluconate in Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-201
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — disulfiram-copper; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DSF-Cu (Experimental): Disulfiram/copper (oral capsules) dosed 80 mg/1.5 mg three times a day for approximately 6 months.
  Interventions: Drug: Disulfiram/Copper; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Disulfiram/Copper — Disulfiram/copper gluconate is taken three times a day.
Drug: Temozolomide (TMZ) — TMZ is given per standard of care

SUMMARY:
This study of DSF-Cu in combination with TMZ for recurrent GBM will evaluate the antitumor effect in patients who have recurrent GBM. Patients will take DSF-Cu daily during their routine standard of care with TMZ therapy for approximately 6 months. Patients will be evaluated for response every 8 weeks. Patients will be followed up 2 years after the last dose of DSF-Cu.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM (WHO grade IV).
* The subject must have completed RT with concurrent TMZ at least 12 weeks prior to the planned start of treatment on this study UNLESS there is pathological verification of recurrent tumor and at least 4 weeks have elapsed since the end of RT with concurrent TMZ.
* Experienced first unequivocal progression of tumor by magnetic resonance imaging (MRI) [as assessed via Radiologic Assessment in Neuro-Oncology (RANO) criteria within 3 months from the last dose of TMZ.
* Karnofsky performance status (KPS) of at least 60%.
* Willing to remain abstinent from consuming alcohol.
* Recovered from the toxic effects of prior therapy to < grade 2 toxicity per NCI CTCAE prior to study registration (except lymphopenia).
* Meets laboratory criteria for the following parameters: ANC, platelets, hemoglobin, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, BUN and creatinine.
* 11. Females of childbearing potential must be willing to use an acceptable method of birth control (i.e., intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.

Exclusion Criteria:

* Radiographic evidence of leptomeningeal dissemination, gliomatosis cerebri, infratentorial tumor, or disease at sites remote from the supratentorial brain.
* Enrolled in another clinical trial testing a novel therapy or drug within the past 4 weeks.
* Received more than one course of radiation therapy or more than a total dose of 75 Gy.
* History of allergic reaction/hypersensitivity to temozolomide, dacarbazine, DSF or Cu.
* Treatment with the following medications are contraindicated with DSF: metronidazole, isoniazid, dronabinol, carbocisteine, lopinavir, paraldehyde, ritonavir, sertraline, tindazole, tizanidine, atazanavir.
* Fever within 3 days prior to study enrollment.
* Active or severe hepatic or renal disease.
* Grade 2 or higher peripheral neuropathy or ataxia per NCI CTCAE
* History of idiopathic seizure disorder schizophrenia, or psychosis unrelated to glioblastoma, corticosteroid, or anti-epileptic medications.
* History of Wilson's disease.
* History of hemochromatosis.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, MD, Study Chair — Washington University School of Medicine in St. Louis
Locations (8):
- United States (8):
  - Beaumont Hospital, Royal Oak, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Lenox Hill Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Huang J, Chaudhary R, Cohen AL, Fink K, Goldlust S, Boockvar J, Chinnaiyan P, Wan L, Marcus S, Campian JL. A multicenter phase II study of temozolomide plus disulfiram and copper for recurrent temozolomide-resistant glioblastoma. J Neurooncol. 2019 May;142(3):537-544. doi: 10.1007/s11060-019-03125-y. Epub 2019 Feb 15. PMID 30771200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSF-Cu
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Disulfiram and Copper Gluconate: Disulfiram/copper (oral capsules) dosed 80 mg/1.5 mg three times a day for approximately 6 months.
  Disulfiram/Copper: Disulfiram/copper gluconate is taken three times a day.
  Temozolomide (TMZ): TMZ is given per standard of care
Arm/Group | Disulfiram and Copper Gluconate
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 61 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21
  Black | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR will be defined as the percentage of patients with complete response (CR) or partial response (PR) according to the RANO criteria.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | DSF-Cu
Number analyzed (Participants) | 21
Participants
  Complete response | 0
  Partial Response | 0

2. Secondary Outcome: Progression Free Survival
Description: Percentage of patients that are free from progressive disease per RANO criteria
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DSF-Cu
Number analyzed (Participants) | 21
percentage of participants | 14 [0 to 28]

3. Secondary Outcome: Overall Survival
Description: Percentage of patients that are alive
Time Frame: 6 months and 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DSF-Cu
Number analyzed (Participants) | 21
percentage of participants
  6 months | 61 [41 to 81]
  12 months | 35 [15 to 54]

4. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of Participants with Grade 3 and 4 serious adverse events
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | DSF-Cu
Number analyzed (Participants) | 23
Participants | 2

5. Secondary Outcome: Median Progression Free Survival
Description: Duration of progression free survival according to RANO criteria
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DSF-Cu
Number analyzed (Participants) | 21
months | 1.7 [1.4 to 1.9]

6. Secondary Outcome: Median Duration of Overall Survival
Description: Duration of overall survival for patients that are alive
Time Frame: 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DSF-Cu
Number analyzed (Participants) | 21
months | 7.1 [5.8 to 8.5]

ADVERSE EVENTS:
Time Frame: 14 months
Groups:
- Group A: Eligible patients must have progressed after standard chemoradiotherapy and within 3 months of the last dose of TMZ.
Arm/Group | Group A
All-Cause Mortality (participants affected / at risk) | 14/23
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=23)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) — Liver enzyme elevation
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03034135/Prot_SAP_001.pdf